CLINICAL TRIAL: NCT07307014
Title: Quick Relief or Real Response? Acute Effects of Percussion Massage Versus Sham Treatment in Individuals With Nonspecific Neck Pain: A Randomized Controlled Trial
Brief Title: Acute Effects of Percussion Massage in Nonspecific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ertugrul Safran, Asst.Prof, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVUçes
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain Musculoskeletal
Keywords: nonspesific neck pain; percussive massage; musculoskeletal disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussion Massage Therapy (Experimental): Participants in this group receive a single session of percussion massage therapy applied to the bilateral upper trapezius muscles.
  Interventions: Device: Percussion Massage Therapy
- Sham Percussion Therapy (Sham Comparator): Participants in this group receive a sham percussion intervention designed to mimic the active treatment without providing mechanical tissue stimulation.
  Interventions: Device: Sham Percussion Therapy

INTERVENTIONS:
Device: Percussion Massage Therapy — Percussion massage therapy is applied using a handheld percussive massage device. The intervention is performed with the participant in a seated position and targets the bilateral upper trapezius muscles for a total duration of 6 minutes. A circular massage head is used to deliver percussive stimulation along the muscle for 2 minutes on each side, followed by focused stimulation at two trigger points using a bullet head attachment for 30 seconds per point at a frequency of 30 Hz.
  Arms: Percussion Massage Therapy
Device: Sham Percussion Therapy — The same percussive massage device is activated to produce comparable sound and vibration cues but is held at a fixed distance from the skin without physical contact. The duration of the procedure and therapist-participant interaction are matched to the experimental intervention to maintain participant blinding.
  Arms: Sham Percussion Therapy

SUMMARY:
This randomized controlled trial aimed to investigate the acute effects of percussion massage therapy compared with a sham intervention on cervical range of motion and pressure pain threshold in individuals with nonspecific neck pain.

DETAILED DESCRIPTION:
Nonspecific neck pain is a common musculoskeletal condition associated with reduced cervical mobility and increased pain sensitivity. Percussion massage therapy has gained popularity as a therapeutic modality; however, evidence regarding its true physiological effects remains limited.

This single-blind randomized controlled trial investigated the immediate effects of percussion massage therapy compared with a sham intervention in individuals with nonspecific neck pain. Participants were randomly allocated to either a percussion massage therapy group or a sham percussion therapy group. Cervical range of motion and pressure pain threshold were assessed before and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria

Adults aged 18 to 60 years

Diagnosis of nonspecific neck pain

Resting neck pain intensity of ≥3 on the Visual Analog Scale (VAS)

Willingness to participate and provide written informed consent

Exclusion Criteria

History of cervical spine fracture, tumor, or inflammatory disease

Previous surgery involving the neck or shoulder region

Neurological deficits related to the cervical spine

Pregnancy or suspected pregnancy

Cognitive impairment or inability to understand study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion (ROM) | Immediately before and immediately after the intervention
  Cervical range of motion (ROM) is assessed in flexion, extension, right and left lateral flexion, and right and left rotation using a digital goniometer. Measurements are performed in a seated position by a blinded assessor following standardized procedures.

SECONDARY OUTCOMES:
Pressure Pain Threshold (PPT) | Immediately before and immediately after the intervention
  Pressure pain threshold (PPT) is measured bilaterally at two standardized points over the upper trapezius muscle using a digital pressure algometer. Pressure is gradually increased until the participant first perceives pain, and the mean of three measurements at each site is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data supporting the findings of this study are available from the corresponding author upon reasonable request. Owing to ethical and privacy considerations, the data were not publicly available